CLINICAL TRIAL: NCT00634023
Title: A Cross-Sectional, Canadian, Multi-Centre Study of Symptom Burden and Clinical Management in Subjects With Gastroesophageal Reflux Disease (GERD) RANGE: Retrospective ANalysis of GErd
Brief Title: Canadian, Multi-Centre Study of Symptom Burden and Clinical Management in Subjects With GERD
Acronym: RANGE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: D9612L00113
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2009-03

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a cross-sectional study of symptom burden and clinical management. A subset of patients who have attended the Primary Care (PC) office with reflux symptoms during a retrospective period of 4 months (Index Visit) are invited to complete health survey questionnaires and partake in a subject-physician/study nurse interview (Visit 1), in order to assess the type, intensity and frequency of GERD symptoms at both visits and describe the treatment provided. Additionally, the impact of GERD on subjects' life, productivity and willingness to pay for GERD symptom relief will be explored. This design will give a "real-life" clinical practice picture in a representative population of PC doctors and subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Ability to complete PRO instruments (non-applicable to "non-attendees")
* Subject with GERD symptom(s). At least presence of troublesome heartburn and/or regurgitation even if not specifically recorded at the Index Visit.
* At least one visit during the Retrospective Visit Period (-6 to -2 months prior to study start).

In the reasons for the Index Visit section of the medical record mention of acid regurgitation and/or heartburn symptom(s) or GERD diagnosis or GERD complications has to be explicit or a treatment decision (prescription) in a previously diagnosed subject although no mention of symptoms is made.

Exclusion Criteria:

* Prophylactic PPI use to reduce the risk of ulcers in subjects being treated with NSAIDs
* PPI treatment to heal an ulcer induced by NSAID treatment
* PPI treatment for H-pylori eradication
* Participation in any other clinical study in the time window between the Index Visit and Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects attending PC offices with reflux symptoms. Subjects must not have participated in any other clinical study in the time window between the Index Visit and Visit 1.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To describe the impact of reflux symptoms on subjects' daily life | Assessed by means of the patient reported outcomes (PROs)

SECONDARY OUTCOMES:
To describe the impact of reflux symptoms on work productivity | Assessed by means of the patient reported outcomes (PROs)

CONTACTS AND LOCATIONS:
Locations (15):
- Canada (15):
  - Research Site, Edmonton, Alberta
  - Research Site, Spruce Grove, Alberta
  - Research Site, North Vancouver, British Columbia
  - Research Site, Windsor, Nova Scotia
  - Research Site, Cornwall, Ontario
  - Research Site, Exeter, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Kanata, Ontario
  - Research Site, London, Ontario
  - Research Site, Nepean, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, North Bay, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, St. Catharines, Ontario
  - Research Site, Woodstock, Ontario